CLINICAL TRIAL: NCT06863194
Title: Effects of Probiotic Supplementation on Disease Progression in Patients With Moderate to Severe Chronic Kidney Disease: A Randomized Controlled Trial
Brief Title: Probiotic Supplementation and Disease Progression in CKD: A Randomized Trial
Acronym: PRO-CKD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Samar Elshahat Saleh, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD.24.06.864
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Kidney Disease, Chronic; Renal Insufficiency, Chronic; Gut Dysbiosis; Uremic Toxins
Keywords: Chronic Kidney Disease (CKD); Probiotics; Gut Microbiota; Uremic Toxins; Indoxyl Sulfate (IS); Inflammation in CKD; Dysbiosis in CKD; Lactobacillus plantarum
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Intervention Group) Arm Title: Probiotic Supplementation Group Description: Participants in t (Experimental): Participants in this group will receive Lactogemikan (Probiotic Supplement), which contains 10 billion CFU of Lactobacillus plantarum per tablet. They will take one tablet daily for 6 months.
  The purpose of this intervention is to evaluate whether probiotic supplementation can slow the progression of chronic kidney disease (CKD) by modulating gut microbiota, reducing systemic inflammation, and decreasing uremic toxin levels.
  Participants will be monitored through clinical visits and laboratory tests at baseline, and 6 months to assess kidney function (eGFR, serum creatinine, urinary protein levels), inflammatory markers (CRP, ferritin, albumin), and gut microbiota composition (urinary indican levels).
  Interventions: Drug: Probiotic Supplementation (Lactobacillus plantarum)
- Arm 2 (Control Group) Arm Title: Placebo Group Description: Participants in this group will receive (Placebo Comparator): Participants in this group will receive a placebo tablet that is identical in appearance, taste, and packaging to the probiotic supplement but contains no active probiotic ingredients. They will take one tablet daily for 6 months.
  This group serves as a control to compare the effects of probiotic supplementation against a non-active intervention. Participants will undergo the same clinical visits and laboratory assessments as the intervention group at baseline, and 6 months.
  Outcomes assessed will include kidney function (eGFR, serum creatinine, urinary protein levels), systemic inflammation markers (CRP, ferritin, albumin), and gut microbiota composition (urinary indican levels) to determine whether the probiotic has a measurable impact compared to the placebo.

INTERVENTIONS:
Drug: Probiotic Supplementation (Lactobacillus plantarum) — Participants in this group will receive Lactogemikan (Probiotic Supplement), which contains 10 billion CFU of Lactobacillus plantarum per tablet. The dose is one tablet daily for 6 months.
  This probiotic is intended to modulate gut microbiota, reduce systemic inflammation, and decrease uremic toxins (indoxyl sulfate) in CKD patients. The intervention will be compared to a placebo to evaluate its effectiveness in slowing CKD progression and improving metabolic and inflammatory markers.
  Arms: Arm 1 (Intervention Group) Arm Title: Probiotic Supplementation Group Description: Participants in t
Drug: Placebo Tablets — Participants in this group will receive an inert placebo tablet that is identical in appearance, taste, and packaging to the probiotic supplement but contains no active probiotic ingredients. The dose is one tablet daily for 6 months.
  The placebo serves as a control to compare the effects of the probiotic intervention. Both groups will undergo identical monitoring and follow-up assessments to determine whether the probiotic has a significant effect on kidney function, inflammation, and gut microbiota composition.

SUMMARY:
The goal of this clinical trial is to learn whether probiotic supplementation can slow disease progression in patients with moderate to severe chronic kidney disease (CKD). The trial will also assess the safety of probiotics in these patients.

The main questions the study aims to answer are:

Does probiotic supplementation improve kidney function by reducing serum creatinine levels and protein in urine? Does it reduce inflammation and metabolic imbalances in CKD patients? Does it affect gut microbiota composition and lower harmful toxins in the body? Is probiotic supplementation safe and well-tolerated in CKD patients?

Participants will:

Be randomly assigned to receive either probiotics or a placebo for 6 months. Have clinic visits every 6 months for checkups, blood tests, and urine tests. Be monitored for any side effects and changes in kidney function. Researchers will compare the probiotic group to the placebo group to determine whether probiotics are effective in slowing CKD progression.

DETAILED DESCRIPTION:
Background & Rationale:

Chronic Kidney Disease (CKD) is associated with significant alterations in gut microbiota, leading to the production and accumulation of uremic toxins such as indoxyl sulfate (IS) and p-cresyl sulfate (PCS). These toxins contribute to systemic inflammation, oxidative stress, and accelerated kidney disease progression, ultimately increasing cardiovascular mortality. The disruption of gut barrier function and dysbiosis are major contributing factors in CKD pathophysiology.

Probiotic supplementation has been proposed as an adjuvant therapy to modulate gut microbiota, enhance intestinal barrier integrity, and reduce systemic inflammation. Probiotics, particularly Lactobacillus species, have been shown to ferment dietary fiber, produce beneficial metabolites, and competitively inhibit harmful bacteria. Despite some promising findings, prior clinical trials have reported inconsistent results, necessitating further investigation into the efficacy of probiotics in slowing CKD progression.

This randomized, double-blind, placebo-controlled clinical trial aims to assess the impact of probiotic supplementation on renal function, systemic inflammation, and gut-derived uremic toxins in patients with moderate to severe CKD (Stages III-IV).

Study Design & Methodology This trial is a parallel-group, double-blind, randomized controlled study with a 1:1 allocation ratio. Participants will be recruited from the Urology and Nephrology Center, Mansoura University, and randomized into either the probiotic intervention group or the placebo control group.

Intervention Details:

Study Group: Participants will receive probiotic supplementation (Lactogemikan; Pescado Pharmaceuticals, Egypt), containing 10 billion CFU of Lactobacillus plantarum per tablet. The dose will be one tablet daily for 6 months.

Control Group: Participants will receive an identical placebo tablet for 6 months.

Both groups will be followed up for an additional 6 months after treatment cessation to evaluate any persistent effects of probiotic supplementation.

Primary & Secondary Outcomes:

The trial will measure:

Primary Outcomes:

Changes in serum creatinine, estimated glomerular filtration rate (eGFR), and urinary protein levels over 12 months.

Secondary Outcomes:

Changes in systemic inflammatory markers (C-reactive protein, ferritin, total cholesterol, albumin).

Alterations in gut microbiota composition, assessed by urinary indican (indoxyl sulfate) levels before and after treatment.

Evaluation of safety and tolerability of probiotic supplementation in CKD patients.

Randomization & Blinding:

Randomization: Conducted via a computerized random sequence generator.

Blinding:

Double-blinded (both participants and investigators are blinded to group assignments).

The probiotic and placebo tablets are identical in appearance, taste, and packaging.

Follow-Up & Monitoring:

Participants will be evaluated at three time points:

Baseline assessment (before treatment initiation) 6-month follow-up (after completing treatment) 12-month follow-up (6 months post-treatment cessation) At each visit, clinical, biochemical, and microbiota assessments will be conducted. Any adverse events will be documented.

Statistical Analysis Plan Data will be analyzed using R statistical software (R Core Team, 2023).

Descriptive statistics will summarize baseline characteristics. Continuous variables will be assessed using the Shapiro-Wilk test for normality.

Depending on normality:

Welch's t-test (normally distributed variables) Mann-Whitney U test (non-normally distributed variables) Categorical variables will be analyzed using the Chi-square test. A p-value < 0.05 will be considered statistically significant. Ethical Considerations & Regulatory Compliance Ethical Approval: The study has been approved by the Institutional Review Board (IRB) of Mansoura Faculty of Medicine, Mansoura University (IRB Code: MD.24.06.864).

Informed Consent: All participants will provide written informed consent before enrollment.

Adverse Events Reporting: Any serious adverse events (SAEs) will be immediately reported to the IRB and Ethics Committee.

Confidentiality: Participant data will be anonymized and stored securely. Significance of the Study This study aims to provide new insights into the therapeutic role of probiotics in CKD patients. If effective, probiotic supplementation may offer a low-cost, non-invasive adjunct therapy to slow kidney disease progression, reduce inflammation, and improve metabolic health.

By investigating the mechanistic role of probiotics in modulating gut-derived toxins, this trial may contribute to developing novel microbiome-targeted interventions in nephrology practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years (both males and females).
* Diagnosed with Chronic Kidney Disease (CKD) Stage III or IV, confirmed by eGFR.
* Stable medical condition with no recent hospitalization for acute kidney injury or other serious illnesses.
* Not currently on probiotic supplementation or prebiotic therapy.
* Willing to provide informed consent and comply with the study protocol, including clinic visits and sample collection.

Exclusion Criteria:

* CKD Stage I, II, or V, or on dialysis.
* Currently using probiotics or prebiotics as part of their diet or treatment.
* History of active malignancy (cancer) or undergoing chemotherapy.
* Significant gastrointestinal disease (e.g., inflammatory bowel disease, irritable bowel syndrome, or recent GI surgery).
* Pregnant or breastfeeding women (due to safety concerns).
* Patients with autoimmune diseases (e.g., lupus, rheumatoid arthritis).
* Individuals on long-term antibiotic or anti-inflammatory medication that could interfere with microbiota composition.
* Individuals with severe behavioral or cognitive disorders that may prevent adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline, and 6 months
  eGFR will be calculated using the CKD-EPI 2021 equation to assess changes in kidney function over time. A slower decline in eGFR in the probiotic group compared to the placebo group would indicate a beneficial effect.

SECONDARY OUTCOMES:
Change in Gut-Derived Uremic Toxins (Indoxyl Sulfate) | Baseline, and 6 months
  Urinary indican (indoxyl sulfate) levels will be measured to assess whether probiotics alter gut microbiota composition and reduce uremic toxin production.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality and ethical considerations, individual participant data (IPD) will not be shared.

REFERENCES:
- [Background] Seth A, Yan F, Polk DB, Rao RK. Probiotics ameliorate the hydrogen peroxide-induced epithelial barrier disruption by a PKC- and MAP kinase-dependent mechanism. Am J Physiol Gastrointest Liver Physiol. 2008 Apr;294(4):G1060-9. doi: 10.1152/ajpgi.00202.2007. Epub 2008 Feb 21. PMID 18292183
- [Background] de Araujo EMR, Meneses GC, Carioca AAF, Martins AMC, Daher EF, Silva Junior GB. Use of probiotics in patients with chronic kidney disease on hemodialysis: a randomized clinical trial. J Bras Nefrol. 2023 Apr-Jun;45(2):152-161. doi: 10.1590/2175-8239-JBN-2022-0021en. PMID 36112723
- [Background] Miranda Alatriste PV, Urbina Arronte R, Gomez Espinosa CO, Espinosa Cuevas Mde L. Effect of probiotics on human blood urea levels in patients with chronic renal failure. Nutr Hosp. 2014 Mar 1;29(3):582-90. doi: 10.3305/nh.2014.29.3.7179. PMID 24559003
- [Background] Tian N, Li L, Ng JK, Li PK. The Potential Benefits and Controversies of Probiotics Use in Patients at Different Stages of Chronic Kidney Disease. Nutrients. 2022 Sep 29;14(19):4044. doi: 10.3390/nu14194044. PMID 36235699